CLINICAL TRIAL: NCT00546312
Title: A Clinical Study Evaluating Use of the Thoracic EXCLUDER Endoprosthesis in the Treatment of Descending Thoracic Aortic Diseases
Brief Title: Clinical Study of Thoracic Excluder Endoprosthesis to Treat Descending Thoracic Aortic Diseases
Acronym: Gore Thoracic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arizona Heart Institute (Other)
Responsible Party: Edward B. Diethrich, MD, Arizona Heart Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G990299
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2009-05

CONDITIONS: Descending Thoracic Aortic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Thoracic EXCLUDER Endoprosthesis — Stent-graft endoprosthesis is inserted by Delivery System via a surgical cutdown (e.g., external iliac artery, femoral artery, common iliac artery conduit, etc.) approach. The insertion method depends on each patient's anatomy and is determined by the Clinical Investigator.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of endovascular repair, using the Thoracic EXCLUDER Endoprosthesis, when used in the treatment of descending thoracic aortic disease as indicated by radiological testing at time of discharge, and 1, 6, 12 months and annually following implantation, and to determine the proportion of patients who experience adverse events during and after the implantation procedure, including disease-specific and overall mortality rates.

DETAILED DESCRIPTION:
Thoracic aortic aneurysm, while relatively rare, is a potentially lethal disorder with a poor long-term prognosis if not treated. As the aortic diameter increases, wall tension becomes higher, leading to further expansion of the aneurysm. Consequently, this disease process is a "progressive and self propagating" phenomena, and the natural history of the disease is progressive expansion of the aneurysm with eventual rupture. Patients with descending thoracic aortic aneurysms frequently have concomitant major medical conditions, making them poor candidates for major surgical procedures. Concomitant conditions may include: hypertension, chronic obstructive pulmonary disease, congestive heart failure, and peripheral vascular disease, including abdominal aortic aneurysm, previous stroke and peripheral arterial occlusive disease.

The accepted treatment for aneurysms deemed to warrant intervention is surgical resection and repair. Operative and post operative complications contributing to early mortality after surgical repair of descending thoracic aortic aneurysms include low cardiac output, pulmonary insufficiency, myocardial infarction, postoperative hemorrhage, pulmonary embolism and sepsis.

In addition to mortality, two of the gravest complications of this surgical procedure, neurologic complications due to spinal cord ischemia, such as paraplegia and paraparesis, and renal failure or dysfunction, remain common.

Dissections, another disease process of the descending thoracic aorta, are rare. Aortic dissections are thought to start with a tear or disruption of the intimal lining of the aorta, either due to medial degenerative diseases, trauma or rupture of an ulcerated intimal plaque. Blood at systemic arterial pressures invades the underlying medial layer of the aortic wall, dissecting the layers of the aortic wall, and forming a false lumen. The dissection then propagates for varying distances and in varying directions along the length of the aorta.

As the false lumen increases in size, arterial flow to the true aortic lumen and to arteries arising from the aorta may be blocked or disrupted. Depending upon the location of the primary intimal tear and the direction of dissection propagation, various vital organs may loose arterial blood supply, and the aorta may rupture into the pericardial sac or pleural space, leading to cardiac tamponade or free pleural rupture. Blood flow from the false lumen may reenter the true lumen through another intimal tear, which may occur proximal or distal to the first, depending on the direction of dissection propagation.

Medical therapy is the first line treatment for dissections of the descending thoracic aorta, and is aimed at reducing the mean, peak and diastolic recoil arterial pressure and the dP/dt while maintaining sufficient pressure to adequately perfuse all vital organs. Surgical intervention is warranted for patients with progression of dissection, impending rupture, refractory hypertension, a sizable localized false aneurysmal component, or continued pain.

A device has been designed to treat disease processes of the descending thoracic aorta. The Thoracic EXCLUDER Endoprosthesis is a device that allows for primary endovascular repair of the descending thoracic aorta and is intended to be used as an intraluminal blood conduit. The Thoracic EXCLUDER Endoprosthesis is a flexible, self-expanding endoprosthesis that is constrained on the leading end of a delivery catheter. A separate balloon catheter, the Thoracic EXCLUDER Balloon Catheter, is used to smooth the endoprosthesis following implantation.

Subjects will undergo an evaluation of the endoprosthesis, and will also be evaluated for device and procedure related adverse events that may have occurred during the follow-up period. Follow-up will be completed at 1, 3, 6, 12, 24, 36, 48, and 60 months. Subject evaluation at 1 and 3 months will include a complete Physical Examination and a CT with contrast enhancement. Subject evaluation at 6, 12, 24, 36, 48, and 60 months will also undergo a complete Physical Examination, a CT with contrast enhancement, and a Chest X-Ray (AP, Lateral, and 2 obliques).

ELIGIBILITY:
Inclusion Criteria:

* Thoracic aortic disease deemed to warrant exclusion in order to prevent rupture or extension including dissection and transections.
* Anatomy meets Thoracic EXCLUDER Endoprosthesis specification criteria.
* Minimum 2 cm non-aneurysmal segment proximal and distal to the aneurysm.

  * < 60 angle in the aortic arch may require additional length of non- aneurysmal segment if the arch is included in the treatment segment.
* The patient is of a "high risk" status for surgical repair. The patient is characterized by the presence of co-morbid factors and/or thoracic aortic pathology that place the patient in a category of prohibitive risk for open repair, and, without intervention, and adverse event could be anticipated within days or weeks. The patient has an ASA score of IV or V.
* Ability to comply with protocol requirements including follow-up.
* Signed Informed Consent Form.

Exclusion Criteria:

* > 4 mm aortic taper and inability to use devices of different diameters, to compensate for the taper, in the treatment area of the aorta.
* Significant thrombus at the proximal or distal implantation sites.
* Planned occlusion of the left carotid or celiac arteries, unless supplemental conduit provided.
* Myocardial infarction within six weeks.
* Degenerative connective tissue disease, e.g. Marfan's or Ehler Danlos Syndrome, unless the proximal and distal implantation sites of the Thoracic EXCLUDER Endoprosthesis are located within previously placed surgical grafts.
* Female of child bearing potential with positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2000-02; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Technical success | following procedure
  Successful completion of the treatment at the initial time of the procedure defined by successful access to the arterial system, deployment, placement and patency of the Thoracic TAG Endoprosthesis at time of procedure.
Treatment Success | 30 days
  Initial technical success and exclusion of the appropriate portion of the descending thoracic aortic disease from the blood circulation, defined as the absence of aneurysm enlargement (if aneurysm present) and avoidance of rupture, without major complications within 30 days of the procedure.
Clinical Success | through 12 months
  Treatment success followed by patency of the graft, and continued exclusion of the appropriate portion of the descending thoracic aortic disease from the blood circulation, without reintervention, rupture, and any major complications through twelve months.

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Diethrich, M.D., Principal Investigator — Arizona Heart Institute
Locations (1):
- Arizona Heart Institute, Phoenix, Arizona, United States

REFERENCES:
- [Background] Fann JI, Miller DC. Endovascular treatment of descending thoracic aortic aneurysms and dissections. Surg Clin North Am. 1999 Jun;79(3):551-74. doi: 10.1016/s0039-6109(05)70024-4. PMID 10410687
- [Background] Bickerstaff LK, Pairolero PC, Hollier LH, Melton LJ, Van Peenen HJ, Cherry KJ, Joyce JW, Lie JT. Thoracic aortic aneurysms: a population-based study. Surgery. 1982 Dec;92(6):1103-8. PMID 7147188
- [Background] Clouse WD, Hallett JW Jr, Schaff HV, Gayari MM, Ilstrup DM, Melton LJ 3rd. Improved prognosis of thoracic aortic aneurysms: a population-based study. JAMA. 1998 Dec 9;280(22):1926-9. doi: 10.1001/jama.280.22.1926. PMID 9851478
- [Background] McNamara JJ, Pressler VM. Natural history of arteriosclerotic thoracic aortic aneurysms. Ann Thorac Surg. 1978 Nov;26(5):468-73. doi: 10.1016/s0003-4975(10)62927-x. PMID 753161
- [Background] Najafi H. 1980: descending aortic aneurysmectomy without adjuncts to avoid ischemia. 1993 update. Ann Thorac Surg. 1993 Apr;55(4):1042-5. doi: 10.1016/0003-4975(93)90150-g. PMID 8466324
- [Background] von Segesser LK, Killer I, Jenni R, Lutz U, Turina MI. Improved distal circulatory support for repair of descending thoracic aortic aneurysms. Ann Thorac Surg. 1993 Dec;56(6):1373-80. doi: 10.1016/0003-4975(93)90684-a. PMID 8267439
- [Background] Hamerlijnck RP, Rutsaert RR, De Geest R, Brutel de la Riviere A, Defauw JJ, Vermeulen FE. Surgical correction of descending thoracic aortic aneurysms under simple aortic cross-clamping. J Vasc Surg. 1989 Apr;9(4):568-73. PMID 2709524
- [Background] Culliford AT, Ayvaliotis B, Shemin R, Colvin SB, Isom OW, Spencer FC. Aneurysms of the descending aorta. Surgical experience in 48 patients. J Thorac Cardiovasc Surg. 1983 Jan;85(1):98-104. PMID 6848892
- [Background] Carlson DE, Karp RB, Kouchoukos NT. Surgical treatment of aneurysms of the descending thoracic aorta: an analysis of 85 patients. Ann Thorac Surg. 1983 Jan;35(1):58-69. doi: 10.1016/s0003-4975(10)61432-4. PMID 6849582
- [Background] Cooley DA, Baldwin RT. Technique of open distal anastomosis for repair of descending thoracic aortic aneurysms. Ann Thorac Surg. 1992 Nov;54(5):932-6. doi: 10.1016/0003-4975(92)90652-k. PMID 1417289
- [Background] Dake MD, Miller DC, Mitchell RS, Semba CP, Moore KA, Sakai T. The
- [Background] Borst HG, Jurmann M, Buhner B, Laas J. Risk of replacement of descending aorta with a standardized left heart bypass technique. J Thorac Cardiovasc Surg. 1994 Jan;107(1):126-32; discussion 132-3. PMID 8283874
- [Background] Lawrie GM, Earle N, De Bakey ME. Evolution of surgical techniques for aneurysms of the descending thoracic aorta: twenty-nine years experience with 659 patients. J Card Surg. 1994 Nov;9(6):648-61. doi: 10.1111/j.1540-8191.1994.tb00899.x. PMID 7841645
- [Background] Laschinger JC, Izumoto H, Kouchoukos NT. Evolving concepts in prevention of spinal cord injury during operations on the descending thoracic and thoracoabdominal aorta. Ann Thorac Surg. 1987 Dec;44(6):667-74. doi: 10.1016/s0003-4975(10)62163-7. PMID 3318742
- [Background] Rutherford RB; editor; Vascular Surgery, Fourth Edition; 1995, W. B. Saunders Co.
- [Background] Bergan JJ, Yao JST; editors; Aneurysms, Diagnosis and Treatment; 1982, Grune and Straton
- [Background] Fann JI, Miller DC. Aortic dissection. Ann Vasc Surg. 1995 May;9(3):311-23. doi: 10.1007/BF02135293. No abstract available. PMID 7632561
- [Background] Torchiana DF, Shin RD, Akins CW, Hilgenberg AD, et. al. Delayed management of traumatic thoracic aortic disruption. Poster abstract presented at the 35th annual meeting of the Society of Thoracic Surgeons, San Antonio, Texas, January 1999
- [Background] Fann JI, Mitchell RS, Dake DC, Miller DC. Results of endovascular stent-grafting in patients with thoracic aortic aneurysm. Progress in Vascular Surgery chapter 19
- [Background] Kato M, Matsuda T, Kaneko M, Kuratani T, Mizushima T, Seo Y, Uchida H, Kichikawa K, Maeda M, Ohnishi K. Outcomes of stent-graft treatment of false lumen in aortic dissection. Circulation. 1998 Nov 10;98(19 Suppl):II305-11; discussion II311-2. PMID 9852919
- [Background] Sacks D, Marinelli DL, Martin LG, Spies JB. Reporting standards for clinical evaluation of new peripheral arterial revascularization devices. Technology Assessment Committee. J Vasc Interv Radiol. 1997 Jan-Feb;8(1 Pt 1):137-49. doi: 10.1016/s1051-0443(97)70530-x. No abstract available. PMID 9025054